CLINICAL TRIAL: NCT05510076
Title: Evaluation of Different Surgical Approaches Used for Conservative Management of Placenta Accreta Spectrum in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdallah Ahmed Refaat, mr., Sohag University
Other Study IDs: Soh-Med-22-08-03
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: in which full-thickness vertical compression suture combined with inflated intrauterine balloon are used to control bleeding
- Group B: in this group, a resective-reconstructive technique is used, which involves resecting the invasive accreta area followed by immediate uterine reconstruction and bladder reinforcement
- Group C: In this group, bilateral uterine artery ligations combined with cervical tamponade which is performed by elevating the cervix into the uterine cavity with Allis forceps, then suturing the anterior and/ or posterior cervical lip(s) into the anterior and/ or posterior uterine segment(s) depending on the site of bleeding with two or three simple interrupted stitches, with the patency of the cervical canal confirmed, followed by closure of the uterine incision

SUMMARY:
The objective of this study is to evaluate different intra-operative procedures to control bleeding in cases of PAS disorders aiming to determine the best procedure regarding maternal morbidity and mortality post-operatively, and to evaluate the long-term effects of conservative management of PAS disorders.

DETAILED DESCRIPTION:
The term "placenta accreta spectrum" (PAS), formerly known as "morbidly adherent placenta" or "abnormally invasive placenta," refers to the aberrant trophoblast invasion of all or a portion of the placenta into the myometrium of the uterus. according to the depth of the villous invasion into the myometrium, the spectrum is assorted into three groups: placenta accreta (villi attach to the myometrium without invading it), placenta increta (villi infiltrate the myometrium), and placenta percreta (villi pierce through the uterine serosa and may infiltrate the surrounding tissues). The optimal strategy for managing PAS disorders remains debatable. Conservative management of PAS disorders includes all techniques aimed at preserving the uterus. Because intraoperative bleeding from PAS disorders is frequently massive and dramatic, causing severe maternal morbidity and mortality, it is essential to have a well-planned, effective, and rapid approach to this surgical challenge.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least one previous caesarean section and suspected PAS disorders by imaging studies

Exclusion Criteria:

* Patients with intraoperative spontaneous placental separation.
* Patients with a preoperative diagnosis of placenta percreta who chose to have an elective hysterectomy.
* Any other associated uterine pathology requiring hysterectomy.
* Coagulation disorders.

Max Age: 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: community sample, any suspected case of PAS disorders.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
successful intervention procedure | 1 day
  Preservation of the uterus
maternal mortality and morbidity | 6 weeks
  ICU admission, need of re-exploration, drop of hemoglobin and hematocrit values, massive blood transfusion, bladder and/ or ureteric injury, coagulopathy, infection and hospital re-admission within 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided